CLINICAL TRIAL: NCT00342368
Title: A Comparison of CPAP Delivered by Helmet and O2 Therapy With a Venturi Mask as First Line Intervention in Early ALI/ARDS
Brief Title: Helmet CPAP vs Venturi O2 to Treat Early ALI/ARDS
Acronym: HelmetCPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prot.pdc181(A.295)/C.E./2004
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: CPAP; ARDS; ALI; Hypoxemia; Intubation
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CPAP through an helmet
  Interventions: Procedure: CPAP delivered by an Helmet
- 2 (No Intervention): O2 therapy with conventional face mask

INTERVENTIONS:
Procedure: CPAP delivered by an Helmet — continuous positive airway pressures delivered through an helmet
  Arms: 1

SUMMARY:
Mechanical ventilation through an endotracheal tube is a lifesaving procedure for acute respiratory failure. However endotracheal intubation increases patient's discomfort and stress, and represents one of the most important predisposing factors for developing nosocomial bacterial pneumonia.

In conscious and cooperative patients non invasive positive pressure ventilation (NPPV) is a safe and effective mean for treating patients with acute respiratory failure (ARF), improving gas exchanges and reducing the rate of complication related to mechanical ventilation. Facial mask, that is the conventional interface for NIV, may induce intolerance because of pain, discomfort or claustrophobia leading to discontinuation of noninvasive ventilation and endotracheal intubation. Thus the improvement of the interface between patient and ventilator seems crucial to achieve a good tolerance allowing the prolonged application of noninvasive ventilation. Attempting to improve tolerability of patients we used a new interface consisting in Helmet made in latex-free PVC.

No prospective randomized controlled study has been published on the comparison between Continuous Positive Airways pressure (CPAP), delivered by an helmet and the medical treatment with Oxygen supplementation to treat early acute respiratory failure and acute lung injury.

Aim of the present protocol is to compare the efficacy of CPAP delivered with helmet and conventional medical treatment with oxygen supplementation via Venturi mask, to prevent ETI in patients with early hypoxemic ARF ( paO2 /FiO2 below 300).

DETAILED DESCRIPTION:
Prevention of Endotracheal Intubation by NIV and CPAP Mechanical ventilation through an endotracheal tube is a lifesaving procedure for acute respiratory failure. However endotracheal intubation increases patient's discomfort and stress, often requiring sedation, may cause injuries of the tracheal mucosa and tracheal stenosis (1), and represents one of the most important predisposing factors for developing nosocomial bacterial pneumonia.

In conscious and cooperative patients non invasive positive pressure ventilation (NPPV) is a safe and effective mean for treating patients with acute respiratory failure (ARF), improving gas exchanges and reducing the rate of complication related to mechanical ventilation .

Noninvasive ventilation and CPAP can be performed by of full face mask. Facial mask may induce intolerance because of pain, discomfort or claustrophobia leading to discontinuation of noninvasive ventilation and endotracheal intubation. During the early phases of hypoxemic acute respiratory failure if disconnection from mechanical ventilation occurs, patients can rapidly deteriorate gas exchanges with potential life threatening consequences. Despite improvements in facial masks characteristics, skin necrosis may occur in 7% of patients treated with NPPV for periods exceeding 72 hours.

Attempting to improve tolerability of patients we used a new interface consisting in Helmet made in latex-free PVC that allows patients to see, read and speech as during noninvasive pressure support ventilation (NPSV) and CPAP ( Continuos Positive Airways Pressure).

The efficacy of a helmet was recently tested and successfully applied to deliver CPAP as out of hospital treatment for patients with pulmonary edema. Recently in a matched controlled study we reported the efficacy of NPPV using the helmet to treat adult patients with hypoxemic ARF in comparison to NPSV using standard facial mask.

No prospective randomized controlled study has been published on the comparison between Continuous Positive Airways pressure (CPAP), delivered by an helmet and the medical treatment with Oxygen supplementation to treat early acute respiratory failure and acute lung injury.

Aim of the present protocol is to compare the efficacy of CPAP delivered with helmet and conventional medical treatment with oxygen supplementation via Venturi mask, to prevent ETI in patients with early hypoxemic ARF ( paO2 /FiO2 less than 300).

Patients enrolled will be randomly assigned to receive either standard treatment with oxygen supplementation delivered by Venturi mask or CPAP through the Helmet. Computer-generated random assignments will be concealed in sealed envelopes The ethic committee of the Catholic University in Rome approved the protocol, and all patients or the next-of-kin will give written informed consent.

Helmet CPAP

During CPAP, the helmet is connected by conventional tubing to a free flow CPAP generator (CaStar Flow generator, Starmed, Italy) with an inspiratory flow more than 45 l/min (Patroniti Intensive Care Med (2003) 29:1680.1687), to avoid the need of a reservoir bag and the risk of rebreathing

The Helmet (CaStar Flow, Starmed, Italy) is made of transparent latex-free PVC that allows patient to see, read and interact with the environment. The helmet is secured by two arm-pit braces at two hooks of the metallic ring that joins the helmet with a seal connection soft collar around the neck. The helmet is available in three different sizes in order to ameliorate comfort and a specific seal connector placed in the metallic ring can be used to allow the passage of a nasogastric tube avoiding air leakage. This connector can be also used to allow patient drinking through a straw. A multiple value PEEP valve ( range 0-20 cm H2O)(Starmed PEEP valve Mirandola Italy) is connected to the expiratory port of the Helmet, where the PEEP value can be confirmed by an anaeroid manometer.

If necessary the helmet can be easily removed and endotracheal intubation can be performed rapidly.

The patients will be not sedated. CPAP will be initiated with a FiO2 equal to or greater than 0.5. PEEP levels will start from 5 cmH2O and augmented by 2 cmH2O stepwise if clinically needed to assure a level of arterial oxygen saturation equal to or greater than 92%.

CPAP level will be reduced progressively on clinical improvement and discontinued if the patient have a PaO2 / FiO2 above 300 and a RR lower than 30 breaths/min, without PEEP and activation of the accessory muscles of respiration

Venturi Mask group Patients assigned to the standard treatment group will receive oxygen supplementation via a Venturi mask starting with a fraction of inspired oxygen equal to or greater than 0.5, and adjusted to achieve an initial level of arterial oxygen saturation equal to or greater than 92%.

Oxygen cessation criteria: the patient with a PaO2 / FiO2 above 300 and a RR lower than 30 breaths/min, without activation of the accessory muscles of respiration

Criteria for endotracheal intubation

Patients failing CPAP or standard treatment will be intubated orotracheally with cuffed endotracheal tubes (internal diameter of 7.5 to 8.5 mm) and mechanically ventilated. Predetermined criteria for endotracheal intubation will be identical for all groups and will include one of the following:

the inability of the patient to tolerate the helmet, including discomfort, claustrophobia or pain.

* PaO2 below 150 and at least, one of the Following
* Loss of alertness or agitation needing sedation
* Signs of exhaustion
* Absence of cough, inability to maintain airway with head in felxion
* Respiratory arrest
* Hemodynamic instability (MAP below 65 mmHg.) frequent recurrent non perfusing dysarrhythmia
* Cardiac arrest
* Signs of patient distress with accessory muscle recruitment and paradoxical abdominal motion
* RR above 35 RR/min
* Respiratory acidosis (pH below 7.3 and PaCO2 above 50 mmHg)

Conventional ventilation after the treatment failure Intravenous benzodiazepines (Midazolam) or propofol will be used for sedation at the moment of intubation, and if possible none of the patients will receive paralyzing agents. The initial ventilator setting will be assist-controlled ventilation mode with a delivered tidal volume of 6-7 ml/kilogram IBW and a initial respiratory rate of 18-25 breaths/min, a PEEP of 5 cmH2O, and a FiO2 of 0.8. Subsequent changes of the ventilator setting will be done according to the NIH protocol. (N Engl J Med 2000;342:1301-8.) All patients will be weaned from the ventilator by reducing the level of pressure support by 4 cmH2O twice and then at 2 hour intervals as tolerated up to 8 cmH2O of pressure support. If the patient will tolerate a pressure support level of 8 cmH2O and an FiO2 of equal to or less than 0.5, a 2 hour T-piece trial will be initiated(11). These patients will be extubated if they maintain a respiratory rate less than 30 breaths/min and a PaO2 greater than 75 mm Hg

Plan of experiment Multicenter, randomized controlled clinical trial. Enrolled patients will be randomly assigned to receive either standard treatment with oxygen supplementation delivered by Venturi mask or CPAP through a Helmet. Each patient will be observed for the following days until discontinuation or failure.

Arterial blood gas levels will be determined at baseline, while breathing through Venturi mask, at 1 hour during CPAP, and at 6-12 hours intervals for the first 24 hours. ABG will be daily determined for the following days until discontinuation or failure.

End Points and Definitions The primary outcome variable will be the evaluation of the need for endotracheal intubation.

Secondary end points will include the improvement of gas exchanges, complications not present on admission (such as ventilator-associated pneumonia or extra-pulmonary sepsis), duration of ventilatory assistance, length of the hospital stay, and ICU mortality. For each patient the number of days free of mechanical ventilation will be recorded during the first 28 days after the admission or until hospital discharge.

Improvement in gas exchange are defined as the ability to increase PaO2:FiO2 ratio above 300 or an increase in this ratio of more than 100 from base line.(4-5) Improvement in gas exchange will be evaluated within 1 hour (initial improvement) after study entry and over time (sustained improvement). Sustained improvement in gas exchange will be defined as ability to maintain the defined improvement in PaO2/FiO2 until mechanical ventilation was discontinued, as confirmed by serial blood gas measurements.

Population of the study Experimental Center This trial is multicenter and involves four different intensive care units in Italy (Università Cattolica del Sacro Cuore, Università dell'Insubria-Varese, Università di Torino, Ospedale S. Gerardo di Monza Power of the study Under the assumptions that the actual difference within the treatment is about 20% (20 vs. 40% intubation rate) with an type 1 error level of 0.05 and with a desired power of 90%, between Helmet and Venturi group, the sample size is computed like 80 in the Helmet group and 80 in the Venturi group. Keeping into account a 20% attrition rate about 190 patient should be enrolled in the study.

The primary end-point will be the proportion of endotracheal intubation in the two groups.

Secondary End-points Secondary end points will be the improvement of gas exchange, complications not present on admission (such as ventilator-associated pneumonia or extra-pulmonary sepsis), complications directly related to noninvasive CPAP as skin breakdown, gastric distension or conjuctivitis, duration of ventilatory assistance, length of the ICU and hospital stay, ICU and 28 days mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acute Hypoxemic Respiratory failure
* Severe Dyspnea at rest
* Pulmonary infiltrates at chest X ray
* PaO2/FiO2<300
* Respiratory Rate > 30 breaths/min

Exclusion Criteria:

* Age < 18 years
* COPD
* CPE
* Patients belonging to Class II-III-IV of the NYHA
* Unstable angina and myocardial infarction/ cardiac surgery within the previous 3 months
* Intubation refused or contraindicated
* Acute Respiratory Acidosis pH < 7.30 and PaCO2 > 50 mmHg
* More than 3 organ failures
* Systolic Pressure < 90 mmHg, under fluid resuscitation or Epinephrine or Norepinephrine > 0.1 gamma/Kg/min
* EKG instability with ventricular arrhythmias
* EXPECTED surgery during the 48 hours following the enrollment
* Coma or seizures
* Decreased level of consciousness (GCS <12)
* Inability to clear secretions
* Pre-defined intubation criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2005-06; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
The number of endotracheal intubations over the study period | period during the ICU stay

SECONDARY OUTCOMES:
The improvement of gas exchange | period during icu stay
The complications not present on admission | period during the icu stay

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, Prof, Study Director — Catholic University of the Sacred Heart
Locations (1):
- UCSC, Policlinico Universitario A. Gemelli, ICU, Rome, Rome, Italy